CLINICAL TRIAL: NCT02289768
Title: Multicentre, Randomized, Parallel, Double-Blind, Vehicle Controlled Study To Evaluate The Efficacy And Safety Of Actikerall® Solution In The Field-Directed Treatment Of Actinic Keratoses Grade I To II (Field Cancerization)
Brief Title: Study To Evaluate The Efficacy And Safety Of Actikerall® Solution In Patients With Grade I-II Actinic Keratoses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Almirall Hermal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 98605101-1401; 2014-001171-31 (EudraCT Number); ALM014 (Other: Almirall Hermal GmbH)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2015-10

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 5-fluorouracil, salicylic acid drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-fluorouracil/salicylic acid (Experimental): Actikerall® solution (5-fluorouracil 0.5%, salicylic acid 10.0%) applied to the affected area once-daily for 12 weeks
  Interventions: Drug: 5-fluorouracil/salicylic acid
- Vehicle (Placebo Comparator): Vehicle solution applied to the affected area once-daily for 12 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: 5-fluorouracil/salicylic acid
  Other Names: Actikerall
  Arms: 5-fluorouracil/salicylic acid
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
The main purpose of this vehicle-controlled study is to determine the efficacy and safety of a solution of Actikerall® (containing 5-fluorouracil 0.5% and salicylic acid 10.0%) in the field-directed treatment of grade I-II actinic keratosis, when it is applied to the affected area once daily for 12 weeks.

A secondary objective of this study is to evaluate the efficacy of Actikerall® solution on subclinical actinic keratosis lesions in a subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant, non-lactating (in the last 3 months) female aged between 18 and 85 years (both inclusive). Women of childbearing potential will follow specific study requirements.
* Patients with at least 4 but not more than 10 clinically confirmed actinic keratoses lesions grade I or II (according to Olsen EA et al. 1991) within a field of cancerization of 25 cm² in the face/forehead or bald scalp.
* Patients with skin type I to IV (according to Fitzpatrick Skin Types)
* Patients free of any significant physical abnormalities (e.g., tattoos, dermatoses) in the potential treatment area that may interfere with area examination or final evaluation.
* Patients in good health condition or free of medical conditions that may interfere with the study results as confirmed by a physical examination, medical history and laboratory analysis.
* Patients who accept to refrain from sunbathing, intense UV-light exposure and the solarium during the study duration.
* Patients willing to stop using moisturizers and topical treatments with anti-aging products, vitamins A, C, and/or E containing ointments and gels and green tea preparations in the treatment area.
* Patients able (physical ability or supportive person) to apply the study preparations correctly and to follow the study procedure and restrictions.
* Patients with at least 3 subclinical lesions in the 25 cm² test area (field) clearly separated from each other and the actinic keratoses lesions (additional inclusion criteria for the patients participating on the sub-clinical lesions sub-study).

Exclusion Criteria:

* Subjects that have received treatment for actinic keratoses within the treatment area in the 3 months previous to Visit 1 (screening).
* Subjects that have received prohibited pharmacological or non-pharmacological treatments for any indication other than actinic keratoses within the treatment area before randomization (Visit 2).
* Subjects that have received prohibited systemic treatments for any indication before randomization (Visit 2).
* Subjects taking phenytoin, methotrexate or sulfonylurea.
* Subjects with dermatological diseases in the treatment area or surrounding area that may be exacerbated by the study treatment or may interfere the study assessments (e.g. psoriasis, eczema).
* Subjects that have currently malignant or benign tumors of the skin within the treatment area (e.g., malignant melanoma, basal cell carcinoma, squamous cell carcinoma).
* Subjects that suffer from any kind of photodermatoses.
* Subjects that have evidence of clinically significant unstable medical conditions.
* Subjects with known hypersensitivity to any of the trial drugs (5-fluorouracil, salicylic acid), to ingredients of the trial formulation, or to drugs of similar chemical classes
* Subjects with allergy against dimethylsulfoxide, ethanol, ethyl acetate, pyroxyline, poly(butyl)methacrylate, and/or methylmethacrylate.
* Subjects with dihydropyrimidine dehydrogenase deficiency (DPD deficiency).
* Subjects that are currently participating or have participated within the 8 weeks prior to Visit 1 in another clinical trial.
* Patients with known drug or alcohol abuse as assessed by the investigator within the 2 years prior to Visit 1.
* Subject is institutionalized because of legal or regulatory order.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete clinical clearance of actinic keratosis lesions in the treatment field | Week 20
  Complete Clinical Clearance is defined as no clinically visible actinic keratosis lesions in the selected treatment area

SECONDARY OUTCOMES:
Percentage of patients with partial clinical clearance of actinic keratosis lesions in the treatment field | Week 20
  Partial clearance is defined as a 75% or greater reduction in the number of clinically visible actinic keratosis lesions in the selected treatment area
Percentage change from baseline in the total number of actinic keratosis lesions | Week 20
Global assessment of efficacy by the physician (Physician Global Assessment) | Week 20
Change from baseline in total score of the Dermatology Life Quality Index (DLQI) | Week 20
Total score of the patients´ treatment satisfaction questionnaire for medication (TSQM) | Week 20
Percentage of patients with complete clearance of three pre-defined subclinical actinic keratosis lesions | Week 20
  Sub-clinical lesions will be determined using reflectance confocal microscopy in a subset of 30 patients
Percentage change from baseline in the three selected actinic keratosis subclinical lesions | Week 20
  Sub-clinical lesions will be determined using reflectance confocal microscopy in a subset of 30 patients
Percentage of patients for which the clearance of one pre-defined representative clinical actinic keratosis lesion is confirmed by reflectance confocal microscopy | Week 20
  Determined using reflectance confocal microscopy in a subset of 30 patients
The number of patients with adverse events | Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Godehard Ocker, Study Director — Almirall Hermal GmbH
Locations (14):
- Germany (10):
  - Almirall Investigational Site #3, Berlin
  - Almirall Investigational Site #5, Berlin
  - Almirall Investigational Site #4, Berlin
  - Almirall Investigational Site #1, Bochum
  - Almirall Investigational Site #8, Bochum
  - Almirall Investigational Site #6, Bonn
  - Almirall Investigational Site #9, Dülmen
  - Almirall Investigational Site #10, Friedrichshafen
  - Almirall Investigational Site #2, Selters
  - Almirall Investigational Site #7, Wuppertal
- United Kingdom (4):
  - Almirall Investigational Site #11, Leicester
  - Almirall Investigational Site #12, Nantwich
  - Almirall Investigational Site #13, Penzance
  - Almirall Investigational Site #14, Penzance

REFERENCES:
- [Derived] Stockfleth E, von Kiedrowski R, Dominicus R, Ryan J, Ellery A, Falques M, Ivanoff N, Azeredo RR. Efficacy and Safety of 5-Fluorouracil 0.5%/Salicylic Acid 10% in the Field-Directed Treatment of Actinic Keratosis: A Phase III, Randomized, Double-Blind, Vehicle-Controlled Trial. Dermatol Ther (Heidelb). 2017 Mar;7(1):81-96. doi: 10.1007/s13555-016-0161-2. Epub 2016 Dec 19. PMID 27995485